CLINICAL TRIAL: NCT00609414
Title: Albumin Use in Burn Patients
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Bruce A. Cairns MD, Department of Surgery, University of North Carolina at Chapel Hill
Other Study IDs: 04-1392
Record Dates: First submitted 2008-01-24; First posted 2008-02-07 (Estimated); Last update posted 2011-04-18 (Estimated); Status verified 2011-04

CONDITIONS: Burns
Keywords: Burns; Albumin; Fluid Resuscitation
MeSH Terms: conditions — Burns

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a study of why and how physicians use albumin during the first 72 hours after a burn injury.

DETAILED DESCRIPTION:
While albumin has been a part of burn resuscitation for many years, its use remains varied and controversial. The purpose of this study is to describe the current practices of albumin administration during the first 72 hours after a burn injury. Participating sites will collect data on patients with at least a 20% Total Body Surface Area (TBSA) burn. Information will be recorded on type and extent of burn injury, basic demographic data, co-morbidities, outcomes and, for the first 72 hours post injury, if albumin was used and why, amount of resuscitation fluids and urine output, and use of vasopressors and diuretics.

Each participating site will retrospectively review 20 charts of consecutive admissions with at least a 20% TBSA burn. In addition, each site will collect data prospectively on 20 more patients with 20% TBSA burns. Prospective data is requested in order to capture as close as possible to "real time" the reasons physicians choose to give albumin. No Protected Health Information (PHI) will be recorded.

Data will be analyzed for patterns of albumin use and reasons for albumin administration.

ELIGIBILITY:
Inclusion Criteria:

* Burn Injury, with and without inhalation injury

Exclusion Criteria:

* <20% Total Body Surface Area Burned
* Comfort care only for the burn injury

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who have 20% and greater Total Body Surface Area burns who received fluid resuscitation for these injuries.
Sampling Method: Non-Probability Sample
Enrollment: 460 (Actual)
Dates: Start 2005-01; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce A. Cairns, MD, Principal Investigator — North Carolina Jaycee Burn Center, University of North Carolina Hospitals
Locations (12):
- United States (11):
  - Arizona Burn Center, Maricopa Medical Center, Phoenix, Arizona
  - Bothin Burn Center, Saint Francis Memorial Hospital, San Francisco, California
  - Shands at the University of Florida Burn Center, Gainesville, Florida
  - Joseph M Still Research Foundation Inc and Doctors Hospital of Augusta, Augusta, Georgia
  - Bothin Burn Center, University of Kansas Hospital, Kansas City, Kansas
  - Regions Hospital Burn Center, Saint Paul, Minnesota
  - North Carolina Jaycee Burn Center, University of North Carolina Hospitals, Chapel Hill, North Carolina
  - Paul and Carol David Foundation Burn Institute, Akron Children's Hospital, Akron, Ohio
  - Shriners Hospitals for Children, Cincinnati, Ohio
  - Oregon Burn Center, Legacy Health System, Portland, Oregon
  - University of Utah Hospitals Burn Center, Salt Lake City, Utah
- Ross Tilley Burn Centre, Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada